CLINICAL TRIAL: NCT05887479
Title: The Effect of Ultrasound-Guided Botulinum Toxin Injections on Pain, Functionality, Spasticity, and Range of Motion in Patients With Post-Stroke Upper Extremity Spasticity
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: insufficient number of patients
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Aylin Ayyıldız, Medical Doctor, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 042023
Record Dates: First submitted 2023-04-09; First posted 2023-06-02 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Cerebrovascular Disorders; Spasticity, Muscle; Botulinum Toxin
MeSH Terms: conditions — Cerebrovascular Disorders; Muscle Spasticity | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Active Comparator): This is the group that will be injected with botulinum toxin for spasticity and stretching exercises will be given.
  Interventions: Drug: Botulinum toxin type A
- Control Group (Placebo Comparator): This is the group that will be injected with %0,9 NaCl for spasticity and stretching exercises will be given.
  Interventions: Drug: %0,9 NaCl

INTERVENTIONS:
Drug: Botulinum toxin type A — Toxin of Clostridium Botulinum
  Arms: Study Group
Drug: %0,9 NaCl — %0,9 NaCl
  Arms: Control Group

SUMMARY:
The patients between the ages of 35-80 who developed spasticity in the upper extremity after stroke will be included.. Botulinum toxin(BT-A) injection will be applied to the study group(n=16) and placebo injection to the control group(n=15) in addition to conventional rehabilitation and stretching exercises. Evaluations will be made before the treatment, in the 2nd week, and in 3rd month after the treatment. Pain relief will be evaluated with the Visual Analog Scale(VAS) and spasticity assessment will be done with the Modified Ashworth Scale(MAS). The functionality will be evaluated with Fugl Meyer Assessment Scale(FMAS) and Box Block Test(BBT).

ELIGIBILITY:
Inclusion Criteria:

* hemiplegia due to a cerebrovascular accident at least 1 month ago
* cognitively competent
* have spasticity of 1 and above according to the Modified Ashworth Scale
* receive at least 3 cubes in the Box Block Test

Exclusion Criteria:

* Patients with upper extremity brachial plexus lesions,
* shoulder subluxation,
* arthritis and joint contracture,
* neglect syndrome,
* cerebellar and brain stem lesions
* those who did not accept the study

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05-25 (Estimated); Primary Completion 2023-07-15 (Estimated); Study Completion 2023-08-15 (Estimated)

PRIMARY OUTCOMES:
Pain - Visual Analog Scale | 2 weeks after treatment
  The shoulder pain of the patients will be evaluated during passive movement of the shoulder joint. The Visual Analogue Scale (VAS), a score between 0 and 10, will be used in the evaluation.
Range of Motion | 2 weeks after treatment
  Passive flexion, abduction and external rotation of the shoulder, supination of the elbow, and extension of the wrist will be evaluated by the same physician by goniometry. In addition, elbow, proximal interphalangeal, and distal interphalangeal joints will be evaluated as a limitation of extension.
Modified Ashworth Scale | 2 weeks after treatment
  The modified Ashworth Scale (MAS) will be used to evaluate spasticity. The adductor, internal rotator of shoulder, flexor of elbow, wrist and finger, pronator of elbow spasticities will be evaluated using MAS while the patient was in the sitting position.
The Fugl-Meyer assessment scale | 2 weeks after treatment
  The Fugl-Meyer assessment scale (FMAS) will be used to evaluate the motor functions of the upper extremity.

SECONDARY OUTCOMES:
Pain - Visual Analog Scale | 3 months after treatment
  The shoulder pain of the patients will be evaluated during passive movement of the shoulder joint. The Visual Analogue Scale (VAS), a score between 0 and 10, will be used in the evaluation.
Range of Motion | 3 months after treatment
  Passive flexion, abduction and external rotation of the shoulder, supination of the elbow, and extension of the wrist will be evaluated by the same physician by goniometry. In addition, elbow, proximal interphalangeal, and distal interphalangeal joints will be evaluated as a limitation of extension.
Modified Ashworth Scale | 3 months after treatment
  The modified Ashworth Scale (MAS) will be used to evaluate spasticity. The adductor, internal rotator of shoulder, flexor of elbow, wrist and finger, pronator of elbow spasticities will be evaluated using MAS while the patient was in the sitting position.
The Fugl-Meyer assessment scale | 3 months after treatment
  The Fugl-Meyer assessment scale (FMAS) will be used to evaluate the motor functions of the upper extremity.